CLINICAL TRIAL: NCT07323966
Title: Feasibility of Mask-Free Radiotherapy for Brain Tumor Patients
Acronym: MASKLESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025/25JUL/316
Record Dates: First submitted 2025-09-24; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Brain Tumor
Keywords: radiotherapy; brain tumor; mask; surface guidance
MeSH Terms: conditions — Brain Neoplasms | interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy session without mask (Experimental): A radiotherapy session without a mask will be simulated twice (during the first week and last week of treatment) during two scheduled treatment sessions.
  Interventions: Device: Surface Guided Radiation Therapy without mask

INTERVENTIONS:
Device: Surface Guided Radiation Therapy without mask — Patients are positioned using SGRT based on the reference position reconstructed from the simulation scanner. They are asked to remain still during the typical duration of a conventional radiotherapy session. Patient motion is monitored by SGRT throughout the simulated session. A CBCT scan is performed before and after the session. No treatment is delivered.

SUMMARY:
The aim of this study is to investigate the technical feasibility of brain radiotherapy without immobilization masks using surface imaging to ensure accurate patient positioning and continuous motion monitoring.

DETAILED DESCRIPTION:
In brain radiotherapy, immobilization using a thermoplastic mask is a standard practice to ensure treatment accuracy. However, this method causes discomfort and anxiety for patients. The development of surface imaging (Surface Guided Radiation Therapy, SGRT) could offer a solution to this problem. SGRT is a non-invasive and non-ionizing imaging technique that uses cameras to capture the patient's position in real-time. In mask-free treatment, the radiation beam can be interrupted when motion exceeds a certain threshold and restarts only when the position is corrected.

Nowadays, very few studies have examined the concept of radiation therapy without immobilization masks using SGRT.

As part of this study, participants will take part in a simulated mask-free session. We will determine the stability of the patient's position in the absence of a mask. Participants will also complete questionnaires concerning their feelings during sessions with and without masks.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Brain tumor treated with fractionated radiotherapy
* Able to read and complete a questionnaire in French

Exclusion Criteria:

* Inability to remain still

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Stability of patient's position | Through the course of radiation therapy (up to 6 weeks)
  The stability of the patient's position will be assessed:
  * on the basis of "internal" movements (of the skull) detected by scanner imaging before and after the simulated session (on-board CBCT)
  * on the basis of surface movements monitored by SGRT throughout the session.

SECONDARY OUTCOMES:
Patient's feelings with and without the mask | Through the course of radiation therapy (up to 6 weeks)
  Patients are asked to fill in a questionnaire about their feelings (comfort, anxiety, claustrophobia, isolation, pain) during radiotherapy sessions with a mask and simulated sessions without an immobilization mask.
Preference of treatment | Through the course of radiation therapy (up to 6 weeks)
  Patients are asked to indicate whether they prefer to be treated with or without a mask.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No